CLINICAL TRIAL: NCT01424007
Title: Diet Composition and Genetics: Effects on Weight, Inflammation and Biomarkers
Brief Title: Metabolism, Exercise and Nutrition at UCSD (MENU Study)
Acronym: MENU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: California Walnut Commission (Other)
Responsible Party: Principal Investigator, Cheryl Rock, Study Principal Investigator, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1U54CA155435-1; 1U54CA155435 (NIH)
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Obese; Nondiabetic
Keywords: Obese; Women; Weight loss; Exercise; Physical activity; Diet; Female
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lower fat diet (Experimental): Participants in this group will be individually counseled and receive print materials on a higher-carbohydrate, lower-fat diet.
  Interventions: Behavioral: Weight loss
- Lower carbohydrate diet (Experimental): Participants in this group will be individually counseled and receive print materials on a lower-carbohydrate, higher-monounsaturated fat diet.
  Interventions: Behavioral: Weight loss
- Walnut-rich diet (Experimental): Participants in this group will be individually counseled and receive print materials on a lower-carbohydrate, walnut-rich higher-fat diet.
  Interventions: Behavioral: Weight loss

INTERVENTIONS:
Behavioral: Weight loss — Participants would receive print materials on diet and exercise and attend group sessions that would meet weekly for the first 4 months, then every two weeks for the next 2 months, and then monthly for the next 6 months over the course of one year.

SUMMARY:
The purpose of the MENU Study is to examine whether there is a differential weight loss response to different dietary macronutrient composition (higher carbohydrate and lower fat versus lower carbohydrate and higher monounsaturated fat [MUFA] or lower carbohydrate and walnut-rich higher fat diets) in a weight loss intervention in healthy obese women, depending on insulin resistance status. Blood samples will be collected to enable analysis of potential mechanisms and differential response across subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 years and older
* Have BMI >30.0 kg/m2 and <40 kg/m2
* Willing and able to participate in clinic visits, group sessions, and telephone and Internet communications at specified intervals
* Able to provide data through questionnaires and by telephone
* Willing to maintain contact with the investigators for 12 months
* Willing to allow blood collections
* No known allergy to tree nuts
* Able to be physically active

Exclusion Criteria:

* Diabetic
* Inability to be moderately physically active
* A history or presence of a comorbid diseases for which diet modification and increased physical activity may be contraindicated
* Currently pregnant/breastfeeding
* Planning to become pregnant within the next year
* Currently enrolled in a weight loss program or diet intervention study
* Current use of weight loss medication or supplements
* Planned surgical procedure that can impact the conduct of the study
* Have plans to relocate from area within the next year
* 6+ months use of meds likely to cause weight gain or prevent weight loss
* Any condition which in the opinion of the investigator makes the subject unsuitable for inclusion in this study

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2011-12; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Weight loss | 1 year
  Weight loss response, depending on insulin status, to diets that differ in macronutrient composition: 1) higher carbohydrate and lower fat, 2) lower carbohydrate and higher monounsaturated fat [MUFA] or 3) lower carbohydrate and walnut-rich higher fat

SECONDARY OUTCOMES:
Blood factors | 1 year
  To examine whether there is a differential response, depending on insulin resistance status, dietary macronutrient composition and weight loss in hormonal factors and markers of inflammation.
Nutrient-gene interactions | 1 year
  To identify nutrient-gene interactions that contribute to differential response of cytokines to weight loss and diet composition.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Rock, PhD, RD, Principal Investigator — University of California, San Diego
Locations (1):
- Moores UCSD Cancer Center, La Jolla, California, United States

REFERENCES:
- [Result] Rock CL, Flatt SW, Pakiz B, Quintana EL, Heath DD, Rana BK, Natarajan L. Effects of diet composition on weight loss, metabolic factors and biomarkers in a 1-year weight loss intervention in obese women examined by baseline insulin resistance status. Metabolism. 2016 Nov;65(11):1605-1613. doi: 10.1016/j.metabol.2016.07.008. Epub 2016 Jul 25. PMID 27733248
- [Result] Le T, Flatt SW, Natarajan L, Pakiz B, Quintana EL, Heath DD, Rana BK, Rock CL. Effects of Diet Composition and Insulin Resistance Status on Plasma Lipid Levels in a Weight Loss Intervention in Women. J Am Heart Assoc. 2016 Jan 25;5(1):e002771. doi: 10.1161/JAHA.115.002771. PMID 26811166
- [Result] Donnan MS, Heath DD, Flatt SW, Pakiz B, Quintana EL, Rana BK, Natarajan L and Rock CL. Factors Associated with Tocopherol Status in Obese Women: Effects of Diet Composition and Weight Loss. Vitam & Miner, 5(3): 147. doi: 10.4172/2376-1318.1000147, 2016.